CLINICAL TRIAL: NCT00464750
Title: The Impact of Temperature of the Injectate on the Precision (Repeatability) of Cardiac Output Measurements Synchronized With the Respiration (the Temperature Study)
Brief Title: Study on the Repeatability of Cardiac Output Measurements Dependence of Temperature of Injectate
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: 4.2006.1012 / NSD15499
Record Dates: First submitted 2007-04-23; First posted 2007-04-24 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-07

CONDITIONS: Heart Diseases
Keywords: Cardiac output; Thermodilution
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Pulmonary artery catheter — Four series of cardiac output measurements, each series consists of eight measurements using cold and eight measurements using tepid injectate. Randomized order of temperature at first series and crossover design.
  Other Names: Baxter

SUMMARY:
This study tests the reliability of thermodilution cardiac output measurements with pulmonary artery catheters in immediate connection with heart surgery. In accordance with our clinical practice, thermal indicator injections are synchronized with respiration. The impact on measurement repeatability of spontaneous vs artificial ventilation and the effect of the injectate temperature is tested.

The study hypothesis is that when injections are synchronized with the respiration, only three injections at room temperature are needed to be within 5 % of the "true" cardiac output in mechanically ventilated patients.

DETAILED DESCRIPTION:
Bolus thermodilution cardiac output measurements by means of a pulmonary artery catheter have been a mainstay of monitoring critically ill patients for more than thirty years. Recent studies have questioned wether the traditional practice of averaging measurements from tree room temperature thermal indicator injections give sufficient precision.

This study tests the number of indicator injections necessary to be within 5 % of the "true" cardiac output (taken as the average of 16 injections) when the injection is synchronized with the respiration. The reliability of the thermodilution measurements are tested A) in sedated, artificially ventilated cardiac surgical patients and B) in the same patients when postoperatively awake and spontaneously breathing. We further compare the use of room temperature and iced thermal indicator injections.

The study hypothesis is that when injections are synchronized with the respiration, only three injections at room temperature are needed to achieve the desired precision in mechanically ventilated patients.

Only patients receiving a pulmonary artery catheter according our institution standard procedure of care will be included.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac surgical patients who receive a pulmonary artery catheter according to the institution clinical criteria -

Exclusion Criteria:

* Acute cardiac surgery
* Preoperative arrythmias

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elective patients for cardiac surgery
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2006-11; Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Idar Kirkeby-Garstad, MD, Ph D, Principal Investigator — St. Olav University Hospital, Trondheim, Norway
Locations (1):
- St Olav University Hospital, Trondheim, Norway

REFERENCES:
- [Result] Kirkeby-Garstad I, Tronnes H, Stenseth R, Sellevold OF, Aadahl P, Skogvoll E. The Precision of Pulmonary Artery Catheter Bolus Thermodilution Cardiac Output Measurements Varies With the Clinical Situation. J Cardiothorac Vasc Anesth. 2015 Aug;29(4):881-8. doi: 10.1053/j.jvca.2014.12.016. Epub 2014 Dec 12. PMID 25976600